CLINICAL TRIAL: NCT02522377
Title: Administration of Subanesthetic Dose of Ketamine and Electroconvulsive Treatment on Alternate Week Days in Patients With Treatment Resistant Depression: A Double Blind Placebo Controlled Trial
Brief Title: Administration of Subanesthetic Dose of Ketamine and Electroconvulsive Treatment for Treatment Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Dr. Murat Altinay, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ketamine ECT
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Severe Depression
Keywords: Ketamine; Electroconvulsive Therapy; Major Depressive Disorder; Treatment Resistant Depression; electroconvulsive treatment; Severe depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Infusions (Experimental): Subjects who are randomized to be on this group will receive a standard dose of ketamine interleaved with Electroconvulsive Treatments.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Subjects who are randomized to be on this group will receive midazolam infusions interleaved with Electroconvulsive Treatments.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — inter venous injections
  Other Names: Ketalar; Calypsol; Ketanest; Tekam
  Arms: Ketamine Infusions
Drug: Midazolam — inter venous injections
  Other Names: Dormicum; Hypnovel; Versed
  Arms: Midazolam

SUMMARY:
In this proof of concept study, the investigators plan to administer iv ketamine interleaved with ECT days.

Patients with treatment resistant depression who are deemed to be eligible for ECT treatment will randomly be assigned to either ketamine or active placebo.

DETAILED DESCRIPTION:
The study will compare the effects of standard ketamine dosing with an active placebo arm.

Hypothesis 1:

The investigators hypothesize that interleaved Electroconvulsive Treatment and active ketamine treatment will lead to a meaningful clinical improvement compared to Electroconvulsive Treatment and placebo treatment arm.

Hypothesis 2:

The investigators hypothesize that interleaved Electroconvulsive Treatment and active ketamine treatment will attenuate cognitive side effects.

Methods and Design:

Patients with treatment resistant depression who are deemed to be eligible for Electroconvulsive Treatment will randomly be assigned to either ketamine or active placebo

Electroconvulsive Treatments:

All patients (independent of their depression scores) will receive the same Electroconvulsive Treatment parameters: Bi-frontal brief pulse (0.5 miliseconds) Electroconvulsive Treatment administered by using Thymatron Electroconvulsive Treatment machine.

Study blinding:

Neither the patients, nor the treating psychiatrist or the nurse will be aware of the patient's assigned arm. The success of blinding will be tested after each ketamine treatment with a questionnaire given to the subject, raters, and treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Males/females at least 18 years of age but no older than 65 years of age
2. Meet Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for Major Depression or Bipolar Disorder, depressed phase, as determined by a clinician's diagnostic evaluation and confirmed by interview using the Mini International Neuropsychiatric Interview (MINI PLUS 5.0.0)
3. A current depressive episode that has lasted a minimum of 4 weeks.
4. Have > 3 trials of antidepressants/augmentation strategies.
5. Have a support system capable of transporting the patient post-treatment.

Exclusion Criteria:

1. Meeting Diagnostic and Statistical Manual of Mental Disorders criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, mental retardation, pervasive developmental disorder.
2. Meeting Diagnostic and Statistical Manual of Mental Disorders criteria for other substance/alcohol dependence within the past 6 months or abuse in the past 3 months.
3. Patients who meet exclusion criteria for ketamine and/or midazolam infusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Altinay, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Center for Behavioral Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with TRD who are admitted to the inpatient psychiatric to receive an acute series of ECT will randomly be assigned to one of the study arms.
Pre-assignment Details: 15 patients with TRD, who were referred to the Cleveland Clinic outpatient depression clinic or ECT service, were recruited in the study. 3 subjects were lost prior to randomization. 2 subjects were lost to follow up after the screening visit, and 1 subject withdrew consent after the baseline visit.12 patients were included in the final analysis.
Groups:
- Ketamine Infusions: Subjects who are randomized to be on this group will receive a standard dose of ketamine alternated with Electroconvulsive Treatments.
  Ketamine: intervenous injections
- Midazolam: Subjects who are randomized to be on this group will receive midazolam infusions interleaved with Electroconvulsive Treatments.
  Midazolam: intervenous injections
Period: Overall Study
Arm/Group | Ketamine Infusions | Midazolam
Started | 7 | 5
Completed | 3 | 5
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Remission Achieved | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine Infusions: Subjects who are randomized to be on this group will receive a standard dose of ketamine interleaved with Electroconvulsive Treatments.
  Ketamine: intervenous injections
- Total: Total of all reporting groups
Arm/Group | Ketamine Infusions | Midazolam | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.9) | 37.6 (15.5) | 38.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 5 | 4 | 9
  Race: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAMD-17) at Last Infusion
Description: Change in HAMD-17 at Infusion 6. Scores range from 0 to 50, with higher scores representing more depression.
Time Frame: visit 17
Population: Analysis was performed on all patients using a mixed effect model. Maximum likelihood estimation allowed for inclusion of all patients, even when loss to follow-up or remission occurred.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
score on a scale | 13.74 (2.62) | 14.97 (2.85)
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority — Superiority test based upon group differences pooled across infusions; p = 0.72, Mixed Models Analysis; Model includes main effect for treatment group and infusion number categorically. Satterthwaite DF=9.987; Mean Difference (Final Values) = 1.22, Standard Error of Mean 3.28 — Midazolam - Ketamine Infusions

2. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) at Last Infusion
Description: Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60
Time Frame: visit 17
Population: Analysis was performed using mixed effect models. Maximum likelihood estimation allowed inclusion of all patients in analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
score on a scale | 22.29 (4.52) | 24.27 (5.93)
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority — Superiority test based upon group differences pooled across infusions in mixed effect model; p = 0.77, Mixed Models Analysis; Model includes main effect for treatment group and infusion number categorically. Satterthwaite DF=7.836; Mean Difference (Final Values) = 1.98, Standard Error of Mean 6.40 — Midazolam - Ketamine Infusions

3. Secondary Outcome: Montreal Cognitive Assessment (MOCA) at Last Infusion
Description: MoCA scores range between 0 and 30. Higher scores reflect higher cognition.
Time Frame: visit 17
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
score on a scale | 24.81 (0.96) | 25.79 (0.97)
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority — Superiority test based upon group differences pooled across infusions; p = 0.40, Mixed Models Analysis; Model includes main effect for treatment group and infusion number categorically. Satterthwaite DF=9.987; Mean Difference (Final Values) = 0.98, Standard Error of Mean 1.12 — Midazolam - Ketamine Infusions

4. Secondary Outcome: Hopkins Verbal Learning Test - Revised (HVLT-R) at Last Infusion
Description: The number of words remembered are recorded. Scores range from 0 to 12 with higher scores reflecting better acquisition.
Time Frame: visit 17
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
score on a scale | 9.42 (0.56) | 11.20 (0.56)
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority — Superiority test based upon group differences pooled across infusions; p = 0.009, Mixed Models Analysis; Model includes main effect for treatment group and infusion number categorically. Satterthwaite DF=9.3634; Mean Difference (Final Values) = 1.78, Standard Error of Mean 0.54 — Midazolam - Ketamine Infusions

5. Secondary Outcome: Controlled Oral Word Association Test (COWAT) at Last Infusion
Description: This is a verbal fluency measure. Outcome is the count of words that meet criteria within 1 minute, so the minimum is 0 and no fixed maximum exists. Higher scores reflect a better outcome.
Time Frame: visit 17
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of words
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
number of words | 33.45 (2.83) | 37.17 (3.03)
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority — Superiority test based upon group differences pooled across infusions; p = 0.34, Mixed Models Analysis; Model includes main effect for treatment group and infusion number categorically. Satterthwaite DF=9.987; Mean Difference (Final Values) = 3.72, Standard Error of Mean 3.71 — Midazolam - Ketamine Infusions

6. Secondary Outcome: Responder Rate on HAMD-17 by Last Infusion
Description: Count of the patients who showed response (>50% decrease).
Time Frame: visit 17
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Infusions | Midazolam
Number analyzed (Participants) | 7 | 5
Participants
  No Response | 4 | 4
  Response | 3 | 1
Statistical Analysis 1: Comparison: Ketamine Infusions vs Midazolam; Test type: Superiority; p = 0.58, Fisher Exact; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.01 to 7.20] — Odds Ratio of Midazolam (numerator) to Ketamine Infusions (denominator)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Ketamine Infusions | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 1/7 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Infusions (N=7) | Midazolam (N=5)
Suicidal Thoughts (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02522377/Prot_SAP_000.pdf